CLINICAL TRIAL: NCT02335931
Title: Follow-up on Cross-sectional Study of Known Population With Charcot Osteoarthropathy - Metabolic, Physiologic and Pathologic Changes
Brief Title: Characterization of the Charcot Foot
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Bo Jansen, MD, Bispebjerg Hospital
Other Study IDs: H-1-2014-055
Record Dates: First submitted 2014-06-27; First posted 2015-01-12 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Charcot's Joint; Complications of Diabetes Mellitus
MeSH Terms: conditions — Arthropathy, Neurogenic; Diabetes Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Frozen full blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Charcot foot: Patients with Charcot foot and diabetes mellitus 1 or 2
- No charcot foot: patients with diabetes mellitus type 1 or 2

SUMMARY:
The project concerns a type of very debilitating diabetic foot complications called Charcots osteoarthropathy (COA). This disease is characterized by a rapidly progressing destruction of the load bearing joints, primarily in the feet, resulting in loss of structure and remodeling. Untreated this cascade leads to the collapse of the bones, meaning severe pain and walking disability for the patient. Reconstruction is often very difficult or impossible, and furthermore the collapse can lead to chronic foot ulcers and infections, which in the worst case can be fatal.

Treatment options are currently limited to early diagnosis and physical offloading (immobilisation), assisted wound healing and surgical intervention.

The purpose of this project is to investigate and describe the bone-related factors, which separate COA from other, less acute, diabetic foot changes. The investigators wish to describe the long term consequences of COA - both anatomically, physiologically and biochemically.

The investigators will be doing this in a follow-up investigations on a group of COA patients tested 8 years ago. Little is known of the long term changes to the bone structure after acute COA, and the investigators want to visualize to what extend the bone damage is permanent.

To do this the investigators will be using DXA-scans, x-ray, blood tests including bone markers, neurophysiological tests and occlusion plethysmography.

DETAILED DESCRIPTION:
please see above

ELIGIBILITY:
Inclusion Criteria:

* Followed in the previous study

Exclusion Criteria:

* Unable to attend follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follow-up study, population of patients referred with charcot foot 8 years ago. Control population without Charcot foot, taken from the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Disease progression in the previously affected foot | initiation

SECONDARY OUTCOMES:
Bone mineral density of os. calcaneus | initiation
Peripheral neuropathy in the feet | initiation
Peripheral blood supply | initiation
Altered levels of bone resorption markers | initiation

OTHER OUTCOMES:
Amputations | initiation
Diabetes regulation | initiation

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus B Jansen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, København NV, Denmark